CLINICAL TRIAL: NCT00847197
Title: A Multicenter, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Lipid-Modifying Effect and Tolerability of MK1903 in Patients With Dyslipidemia
Brief Title: A Study to Evaluate MK1903 in Patients With Dyslipidemia (MK1903-004)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1903-004; 2009_542
Record Dates: First submitted 2009-02-18; First posted 2009-02-19 (Estimated); Results first posted 2010-09-22 (Estimated); Last update posted 2015-12-21 (Estimated); Status verified 2015-11

CONDITIONS: Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — 1a,3,5,5a-tetrahydro-1H-2,3-diazacyclopropa(a)pentalene-4-carboxylic acid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): MK1903
  Interventions: Drug: MK1903
- 2 (Placebo Comparator): Placebo to MK1903
  Interventions: Drug: Comparator: Placebo

INTERVENTIONS:
Drug: MK1903 — Three 50 mg capsules MK1903 by mouth every 8 hours for 4 weeks. All participants will receive placebo for a 2 week run-in period.
  Arms: 1
Drug: Comparator: Placebo — Three 50 mg capsules placebo to MK1903 every 8 hours for 4 weeks. All participants will receive placebo for a 2 week run-in period.
  Arms: 2

SUMMARY:
This study will evaluate the lipid-modifying effect and tolerability of MK1903 when compared to placebo in patients with dyslipidemia who are not on a statin or other lipid-modifying therapy.

ELIGIBILITY:
Inclusion Criteria:

* Participant is not on a statin or other lipid-modifying therapy
* Low or moderate risk participant
* Male participants, and female participants not of reproductive potential

Exclusion Criteria:

* Female participant of reproductive potential
* Participant is pregnant, breastfeeding, or expecting to conceive during the study
* Participant has history of cancer within 5 years of study (except certain types of skin and cervical cancer)
* Participant is a user of recreational or illicit drugs or has a recent history of drug and/or alcohol abuse
* Participant has donated or received blood within 8 weeks of study start or intends to give/receive blood during the study
* Participant consumes more than 3 alcoholic drinks per day or more than 14 alcoholic drinks per week
* Participant is currently experiencing menopausal hot flashes
* Participant currently engages in vigorous exercise or an aggressive diet regimen
* Participant is at high risk for heart conditions
* Participant has Type 1 or Type 2 diabetes mellitus
* Participant has poorly controlled cardiac arrhythmias
* Participant has a history of stroke or other hemorrhage
* Participant has poorly controlled high blood pressure
* Participant has a thyroid condition or other endocrine/metabolic disease that would affect serum lipids
* Participant has a disease of the kidney or liver
* Participant has an ulcer within 3 months of screening
* Participant is Human Immunodeficiency Virus (HIV) positive
* Participant is taking cyclical hormonal contraceptives or non-continuous hormone replacement therapy
* Participant is taking or has taken an Organic Anion Transporter (OAT1/3) inhibitor/substrate within 3 days of screening
* Participant has taken an anti-obesity medication within 3 months of screening
* Participant is taking coumarins
* Participant is taking Non-steroidal Anti-inflammatory Drugs (NSAIDs) (acetaminophen and Cyclooxygenase-2 (COX-2) inhibitors are allowed)
* Participant is taking more than 100 mg aspirin per day
* Participant is being treated with oral, intravenous, or injected corticosteroids or anabolic agents

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2008-06; Primary Completion 2009-09 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited at 26 sites in 8 different countries from February 2009 to August 2009.
Pre-assignment Details: Participants had a 2-week placebo run-in period prior to randomization. 402 participants were screened of which 211 participants were excluded (194 participants did not meet inclusion criteria, 15 participants withdrew, 1 participant was lost to follow-up and 1 participant had an adverse event).
Groups:
- Placebo: Three 50 mg capsules placebo to MK1903 every 8 hours for 4 weeks. All participants will receive placebo for a 2 week run-in period.
Period: Overall Study
Arm/Group | MK1903 | Placebo
Started | 116 | 75
Completed | 92 | 70
Not Completed | 24 | 5
Not completed — Adverse Event | 21 | 3
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK1903 | Placebo | Total
Number analyzed (Participants) | 116 | 75 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (10.4) | 50.9 (11.1) | 51.9 (10.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45 | 28 | 73
  Male | 71 | 47 | 118
Region [Number; unit: participants] — Ex-United States: Malaysia, Canada, Peru, Philipines, Colombia, Sweden, Finland
  participants
    United States | 56 | 38 | 94
    Ex-United States | 60 | 37 | 97
Body Mass Index (BMI) Category [Number; unit: participants]
  < 25 | 20 | 14 | 34
  25 - 30 | 65 | 42 | 107
  31 - 39 | 28 | 17 | 45
  => 40 | 3 | 2 | 5
Coronary Heart Disease (CHD) Risk Category [Number; unit: Participants]
  Low Risk | 90 | 59 | 149
  Multiple Risk | 26 | 16 | 42
Prior Niacin History [Number; unit: Participants]
  Yes | 10 | 11 | 21
  No | 106 | 64 | 170
Glycemic Status [Number; unit: Participants]
  Normal (< 100 mg/dL) | 79 | 53 | 132
  Impaired Fasting Glucose ( ≥ 100 & ≤ 125 mg/dL) | 36 | 21 | 57
  Others (> 125 mg/dL) | 1 | 1 | 2
Weight [Mean (Standard Deviation); unit: Kilogram] | 81.9 (17.9) | 81.6 (17.5) | 81.7 (17.7)
Height [Mean (Standard Deviation); unit: Centimeter] | 168.3 (10.5) | 167.9 (10.2) | 168.2 (10.3)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 28.7 (5.0) | 28.7 (4.5) | 28.7 (4.8)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 122.9 (13.6) | 122.3 (13.5) | 122.7 (13.5)
Diastolic Blood Pressure [Mean (Standard Deviation); unit: mm Hg] | 77.9 (8.9) | 77.1 (9.0) | 77.6 (8.9)
Pulse [Mean (Standard Deviation); unit: beats/minute] | 67.8 (8.8) | 68.5 (8.9) | 68.1 (8.8)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Low-Density Lipoprotein Cholesterol (LDL-C) (mg/dL)
Time Frame: Baseline and Week 4
Population: The Full Analysis Set (FAS) population served as the primary population for the analysis of efficacy data. FAS is a subset of all randomized participants with following reasons for exclusion: 1. failure to receive at least 1 dose of study treatment 2. lack of any post-randomization endpoint data subsequent to at least 1 dose of study treatment.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | MK1903 | Placebo
Number analyzed (Participants) | 112 | 75
Percent Change | -0.3 (16.3) | -1.5 (12.9)
Statistical Analysis 1: Comparison: MK1903 vs Placebo; For the analysis of percent change from baseline in LDL-C at study endpoint, a Longitudinal Analysis of Covariance (ANCOVA) method was used. The repeated measures model included terms for treatment, time (Day 15, 29), and the interaction of time-by-treatment. The analysis model also adjusted for baseline, baseline-by-time interaction, region and gender; Test type: Superiority or Other; p = 0.926, Mixed Models Analysis — The significance test was 2-tailed with α=0.05; The test for the treatment difference in terms of percentage change from baseline to a given time point was done using the contrast statement; Mean Difference (Final Values) = 0.2, 95% CI 2-sided [-3.9 to 4.3], Standard Error of Mean 2.1

2. Primary Outcome: Percent Change From Baseline in High-Density Lipoprotein Cholesterol (HDL-C) (mg/dL)
Time Frame: Baseline and Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | MK1903 | Placebo
Number analyzed (Participants) | 112 | 75
Percent Change | 6.0 (13.0) | 0.7 (11.7)
Statistical Analysis 1: Comparison: MK1903 vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p = 0.013, Mixed Models Analysis — The significance test was 2-tailed with α=0.05; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 4.6, 95% CI 2-sided [1.0 to 8.1], Standard Error of Mean 1.8

3. Secondary Outcome: Percent Change From Baseline in Triglycerides (mg/dL)
Time Frame: Baseline and 4 Weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | MK1903 | Placebo
Number analyzed (Participants) | 112 | 75
Percent Change | -13.2 (32.7) | -2.0 (39.5)
Statistical Analysis 1: Comparison: MK1903 vs Placebo; Triglycerides was analyzed by non-parametric methods with terms for treatment, gender and region. Specifically, the analysis of variance (ANOVA) model was applied to the Tukey's normal scores of the percent change from baseline. The estimate of the difference in medians between MK1903 and the placebo groups utilizing the Hodges-Lehmann estimate and a distribution-free 95% CI for the difference based on Wilcoxon's rank sum test was provided; Test type: Superiority or Other; p = 0.02, Wilcoxon's Rank Sum Test; The significance test was 2-tailed with α=0.05; Median Difference (Final Values) = -10.3, 95% CI 2-sided [-18.9 to -1.9], Standard Error of Mean 8.6

ADVERSE EVENTS:
Time Frame: Reported Adverse Event (AE) data were collected from 6-Feb-09 to 5-Oct-09.
Description: AE information was collected by continuous monitoring of participant's labs and clinical symptoms during the course of the study. AEs were usually reported during routine clinic visits and the 14-day telephone contact conducted after the participant's last visit and the expected date of Visit 4 for discontinued participants.
Arm/Group | MK1903 | Placebo
Serious Adverse Events (participants affected / at risk) | 0/116 | 0/75
Other Adverse Events (participants affected / at risk) | 76/116 | 26/75
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MK1903 (N=116) | Placebo (N=75)
Eye disorders (Eye disorders) | 1 | 2
Gastrointestinal disorders (Gastrointestinal disorders) | 3 | 3
General disorders and administration site conditions (General disorders) | 0 | 4
Infections and infestations (Infections and infestations) | 5 | 4
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 5 | 3
Investigations (Investigations) | 3 | 1
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 4 | 4
Nervous system disorders (Nervous system disorders) | 18 | 5
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 5 | 0
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 32 | 2
Vascular disorders (Vascular disorders) | 42 | 8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.